CLINICAL TRIAL: NCT01229215
Title: A Phase Ib/II, Multicenter, Randomized, Single-Masked, Sham Injection-Controlled Study of Safety, Tolerability, and Evidence of Activity of FCFD4514S Intravitreal Injections Administered Monthly or Every Other Month to Patients With Geographic Atrophy
Brief Title: A Study of Safety, Tolerability, and Evidence of Activity of FCFD4514S Administered Monthly or Every Other Month to Patients With Geographic Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFD4870g; GX01456 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- FCFD4514S (Experimental)
  Interventions: Drug: FCFD4514S
- sham (Sham Comparator)
  Interventions: Drug: sham

INTERVENTIONS:
Drug: FCFD4514S — Repeating intravitreal injection
  Arms: FCFD4514S
Drug: sham — Repeating sham injection
  Arms: sham

SUMMARY:
This is a Phase Ib/II, multicenter, randomized, single-masked, sham-injection-controlled study of safety, tolerability, and evidence of activity of FCFD4514S intravitreal injections administered monthly or every other month in patients with geographic atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide signed Informed Consent; in addition, at U.S. sites, Health Insurance Portability and Accountability Act (HIPAA) authorization, in other countries, as applicable according to national laws
* Well-demarcated area of GA secondary to age-related macular degeneration (AMD) in the absence of choroidal neovascularization (CNV)

Exclusion Criteria:

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation in the study eye
* Prior treatment with Visudyne, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* GA in either eye due to causes other than AMD
* Diabetic retinopathy in either eye
* Active or history of wet AMD in either eye
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or that renders the patient at high risk for treatment complications
* Active malignancy or history of malignancy within the past 5 years
* Previous participation in any studies of investigational drugs within 3 months preceding Day 0

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Growth rate of geographic atrophy (GA) lesion area from baseline | Month 18

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) from baseline | Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Erich Strauss, M.D., Study Director — Genentech, Inc.
Locations (35):
- United States (29):
  - Tucson, Arizona
  - Beverly Hills, California
  - San Francisco, California
  - Santa Barbara, California
  - Torrance, California
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Palm Beach Gardens, Florida
  - Pensacola, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Edina, Minnesota
  - Lynbrook, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - West Columbia, South Carolina
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Dallas, Texas
  - Milwaukee, Wisconsin
- Germany (6):
  - Bonn
  - Freiburg im Breisgau
  - Heidelberg
  - Leipzig
  - Münster
  - Tübingen

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- [Derived] Sivaprasad S, Tschosik E, Kapre A, Varma R, Bressler NM, Kimel M, Dolan C, Silverman D. Reliability and Construct Validity of the NEI VFQ-25 in a Subset of Patients With Geographic Atrophy From the Phase 2 Mahalo Study. Am J Ophthalmol. 2018 Jun;190:1-8. doi: 10.1016/j.ajo.2018.03.006. Epub 2018 Mar 10. PMID 29530781
- [Derived] Kimel M, Leidy NK, Tschosik E, Dolan C, Souied EH, Varma R, Bressler NM. Functional Reading Independence (FRI) Index: A New Patient-Reported Outcome Measure for Patients With Geographic Atrophy. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6298-6304. doi: 10.1167/iovs.16-20361. PMID 27893095
- [Derived] Hariri A, Nittala MG, Sadda SR. Outer retinal tubulation as a predictor of the enlargement amount of geographic atrophy in age-related macular degeneration. Ophthalmology. 2015 Feb;122(2):407-13. doi: 10.1016/j.ophtha.2014.08.035. Epub 2014 Oct 12. PMID 25315664